CLINICAL TRIAL: NCT00495989
Title: The Relationship Between Saliva and Dental Calculus in a Population of Institutionalized Handicapped Persons
Brief Title: Saliva and Dental Calculus in Handicapped People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007/197
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Disabled Persons
Keywords: Handicapped individuals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: saliva sampling + dental calculus collection

SUMMARY:
This is an evaluation of potential differences in saliva composition and dental calculus composition between orally fed and tube fed individuals in an institutional environment.

ELIGIBILITY:
Inclusion Criteria:

* handicapped (mentally and/or physically) persons in an institute
* older than 5 years of age
* both sexes
* full medical records available

Exclusion Criteria:

* healthy individuals
* disabled individuals not staying in an institution

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Saliva composition and dental calculus composition

CONTACTS AND LOCATIONS:
Overall Officials: Johan Aps, DDS, MSc, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be